CLINICAL TRIAL: NCT01682408
Title: An Open-label, Single-center, 2-Part, Randomized Study to Assess the Pharmacokinetics of R406 in Healthy Subjects When Fostamatinib 150 mg is Administered Alone in Fed and Fasted State and in Combination With Ranitidine in Fasted State, and to Assess the Relative Bioavailability of Process Variants of Tablets
Brief Title: Assess Pharmacokinetics of Fostamatinib in Fed and Fasted State in Combination With Ranitidine to Assess Bioavailability
Acronym: PK Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00019
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Pharmacokinetics
Keywords: R406,; Fostamatinib,; Phase I,; Healthy Subjects,; Pharmacokinetics,; Fed/Fasted
MeSH Terms: interventions — Ranitidine

ARMS (5):
- Part A1 (Active Comparator): 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference), fed 3 x 50mg microcrystalline cellulose-based 13% drug loaded tablets,(blue) fed
  Interventions: Drug: Fostamatinib - 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference); Drug: Fostamatinib - 3 x 50mg microcrystalline cellulose-based 13% drug loaded tablets,(blue) fed
- Part A2 (Active Comparator): 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference) 3 x 50mg microcrystalline cellulose-based 13% drug loaded tablets,(blue) fed 150 mg ranitidine
  Interventions: Drug: Fostamatinib - 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference); Drug: Fostamatinib - 3 x 50mg microcrystalline cellulose-based 13% drug loaded tablets,(blue) fed; Drug: Ranitidine
- Part B1 (Active Comparator): 1 x 150mg mannitol based 38% drug-loaded tablet (batch variant A)
  Interventions: Drug: Fostamatinib - 1 x 150mg mannitol based 38% drug-loaded tablet (batch variant A)
- Part B2 (Active Comparator): 1 x 150mg mannitol based 38% drug loaded tablet (batch variant B)
  Interventions: Drug: Fostamatinib - 1 x 150mg mannitol based 38% drug loaded tablet (batch variant B)
- Part B3 (Active Comparator): 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference)
  Interventions: Drug: Fostamatinib - 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference)

INTERVENTIONS:
Drug: Fostamatinib - 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference) — 1 x 150mg mannitol-based 38% drug-loaded tablet(orange reference)
  Arms: Part A1; Part A2; Part B3
Drug: Fostamatinib - 3 x 50mg microcrystalline cellulose-based 13% drug loaded tablets,(blue) fed — 3 x 50mg microcrystalline cellulose-based 13% drug loaded tablets,(blue) fed
  Arms: Part A1; Part A2
Drug: Fostamatinib - 1 x 150mg mannitol based 38% drug-loaded tablet (batch variant A) — 1 x 150mg mannitol based 38% drug-loaded tablet (batch variant A)
  Arms: Part B1
Drug: Fostamatinib - 1 x 150mg mannitol based 38% drug loaded tablet (batch variant B) — 1 x 150mg mannitol based 38% drug loaded tablet(batch variant B)
  Arms: Part B2
Drug: Ranitidine — 150 mg ranitidine
  Arms: Part A2

SUMMARY:
Study to Assess the Pharmacokinetics of R406 in Healthy Subjects when Fostamatinib 150 mg is Administered Alone in Fed and Fasted state and in Combination with Ranitidine in Fasted State, and to Assess the Relative Bioavailability of Process Variants of Tablets

DETAILED DESCRIPTION:
An Open-label, Single-center, 2-Part, Randomized Study to Assess the Pharmacokinetics of R406 in Healthy Subjects when Fostamatinib 150 mg is Administered Alone in Fed and Fasted state and in Combination with Ranitidine in Fasted State, and to Assess the Relative Bioavailability of Process Variants of Tablets

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures including the genetic sampling and analyses
* Volunteers will be males or females aged 18 to 55 years (inclusive) and with a weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2 inclusive.
* Provision of signed, written, and dated informed consent for optional genetic research. If a volunteer declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the volunteer.
* Male volunteers should be willing to use barrier contraception, ie, condoms from the day of first dosing until 2 weeks after dosing with the IP in Treatment Period 5.
* Females must have a negative pregnancy test at screening and on admission to the CPU (including check-in at each treatment period), must not be lactating and must be of non childbearing potential, confirmed at screening

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IP
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics profile of R406 in terms of maximum observed plasma concentration (Cmax) and area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC). | Day 1 (predose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours postdose

SECONDARY OUTCOMES:
Pharmacokinetic profile of R406 in terms of area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-t)], time to Cmax (tmax), terminal half-life (t1/2λz), terminal rate constant (λz). | Day 1 (predose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Description of the safety profile in terms of frequency of adverse events. | up to 3 - 5 days after discharge
Description of the safety profile in terms of severity of adverse events. | up to 3 - 5 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, Principal Investigator — Quintiles Phase I unit 6700 w 115th st Overland Park, Ks 66211; Christopher D O'Brien, MD PHD, Study Director — AstraZeneca
Locations (1):
- Overland Park, Kansas, United States